CLINICAL TRIAL: NCT00046995
Title: 5-Fluorouracil-Leucovorin With or Without Carboplatin as Adjuvant Treatment for Primary Dukes B2-C Colon Cancer; Chronomodulated Versus Standard Administration. A Multicenter Randomized Phase III Trial of the GRECCR-Belgium (Study 03).
Brief Title: Combination Chemotherapy in Treating Patients With Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe Regional d'Etudes du Cancer Colorectal (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000257228; GRECCR-03; EU-20201
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2002-11

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage IIB colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Carboplatin; Fluorouracil; Leucovorin; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: carboplatin
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which schedule of chemotherapy is most effective in treating colon cancer.

PURPOSE: Randomized phase III trial to compare different schedules of chemotherapy using carboplatin with fluorouracil and leucovorin in treating patients who have stage IIB or stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival of patients with completely resected stage IIB or III colon cancer treated with adjuvant chronomodulated vs standard schedule fluorouracil and leucovorin calcium with or without carboplatin.
* Compare the overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Determine the dose intensities of fluorouracil and carboplatin in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and disease stage (IIB vs III). Patients are randomized to 1 of 4 treatment arms.

* Arm I (standard schedule): Patients receive fluorouracil (5-FU) IV continuously and leucovorin calcium (CF) IV on days 1 and 2.
* Arm II (standard + carboplatin schedule): Patients receive 5-FU and CF as in arm I plus carboplatin IV on day 1.
* Arm III (chronomodulated schedule): Patients receive 5-FU IV continuously and CF IV continuously on days 1-4.
* Arm IV (chronomodulated + carboplatin schedule): Patients receive 5-FU and CF as in arm III plus carboplatin IV continuously on days 1-4.

Quality of life is assessed.

Treatment in all arms repeats every 14 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 660-800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon

  * Stage IIB or III (Dukes stage B2 or C)
  * Complete curative resection performed within the past 7 weeks (negative margins)
  * No local or regional relapsed disease
* Tumor more than 15 cm above the anal margin
* Carcinoembryonic antigen less than 5 ng/mL (after surgery)
* No rectal cancer
* No metastatic disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No serious coronary disease

Other

* Not pregnant
* Fertile patients must use effective contraception
* No concurrent infectious disease
* No other malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy (before or after surgery)

Surgery

* See Disease Characteristics

Other

* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2001-05

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Tolerability
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Christian N.J. Focan, MD, PhD, Study Chair — Clinique Saint-Joseph
Locations (2):
- Belgium (2):
  - Centre Hospitalier Hutois, Huy
  - Clinique Saint-Joseph, Liège